CLINICAL TRIAL: NCT05370235
Title: A Proof of Concept, Phase IIa, Open Label Study to Evaluate the Safety and Efficacy of Subcutaneous Implants of Afamelanotide in Patients With Xeroderma Pigmentosum C and V (XPC and XPV)
Brief Title: A Study to Evaluate the Safety and Efficacy of Afamelanotide in Patients With Xeroderma Pigmentosum C and V
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinuvel Europe Limited (Industry)
Responsible Party: Sponsor
Organization: Clinuvel Pharmaceuticals Limited (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CUV152
Record Dates: First submitted 2022-04-21; First posted 2022-05-11 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Xeroderma Pigmentosum
MeSH Terms: conditions — Xeroderma Pigmentosum | interventions — afamelanotide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Afamelanotide (Experimental)
  Interventions: Drug: Afamelanotide

INTERVENTIONS:
Drug: Afamelanotide — Patients will receive afamelanotide every two weeks for twelve weeks and undergo a follow up visit 6 months later.

SUMMARY:
The CUV152 study will evaluate the safety of afamelanotide in XP-C and XP-V patients, as well as the drug's ability to assist reparative processes following ultraviolet (UV) provoked DNA damage of the skin. It will assess whether SCENESSE® increases the amount of UV light needed to cause DNA damage of skin cells, as well as the extent of skin repair before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient with a molecular-genetically confirmed diagnosis of XP-C or XP-V;
* Aged 18-75 years.

Exclusion Criteria:

* Known allergy to afamelanotide or the polymer contained in the implant;
* Presence of severe hepatic disease or hepatic impairment;
* Renal impairment;
* Any other medical condition which may interfere with the study protocol;
* Existing melanoma;
* Female who is pregnant or lactating;
* Females of child-bearing potential (pre-menopausal, not surgically sterile) not using adequate contraceptive measures;
* Sexually active man with a partner of child-bearing potential who is not using adequate contraceptive measures;
* Use of any other prior and concomitant therapy which may interfere with the objective of the study;
* Participation in a clinical trial for an investigational agent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2022-03-28 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in minimal erythema dose (MED) in patients with XP-C. | From baseline to day 76.
  MED is the lowest dose of UV light that causes reddening of the skin.
Change in MED in patients with XP-V. | From baseline to day 76.
  MED is the lowest dose of UV light that causes reddening of the skin.

SECONDARY OUTCOMES:
Changes in UV-induced DNA damage, as assessed by quantification of UV photoproduct levels in patients with XP-C. | From baseline to day 76.
  Analysis of UV photoproducts from skin samples.
Changes in UV-induced DNA damage repair capacity, as assessed by quantification of DNA repair mechanisms in patients with XP-C. | From baseline to day 76.
  Analysis of DNA repair mechanisms from skin samples.
Changes in UV-induced DNA damage, as assessed by quantification of UV photoproduct levels in patients with XP-V. | From baseline to day 76.
  Analysis of UV photoproducts from skin samples.
Changes in UV-induced DNA damage repair capacity, as assessed by quantification of DNA repair mechanisms in patients with XP-V. | From baseline to day 76.
  Analysis of DNA repair mechanisms from skin samples.
Change in skin disease severity in patients with XP-C (A). | From baseline to day 76.
  The higher the score, the more severe the disease.
Change in skin disease severity in patients with XP-V (A) | From baseline to day 76.
  The higher the score, the more severe the disease.
Change in skin disease severity in patients with XP-C (B). | From baseline to day 76.
  The higher the score, the more severe the disease.
Change in skin disease severity in patients with XP-V (B). | From baseline to day 76.
  The higher the score, the more severe the disease.
Change in skin disease severity in patients with XP-C (C). | From baseline to day 76.
  The higher the score, the more severe the disease.
Change in skin disease severity in patients with XP-V (C). | From baseline to day 76.
  The higher the score, the more severe the disease.
Change in quality of life assessed by a disease specific tool (A) in patients with XP-C. | From baseline to day 76.
  Higher scores represent worse health-related quality of life.
Change in quality of life assessed by a disease specific tool (A) in patients with XP-V. | From baseline to day 76.
  Higher scores represent worse health-related quality of life.
Change in quality of life assessed by a validated global quality of life tool (B) in patients with XP-C. | From baseline to day 76.
  Score calculated in impairment percentages, with higher numbers indicating greater impaired quality of life.
Change in quality of life assessed by a validated global quality of life tool (B) in patients with XP-V. | From baseline to day 76.
  Score calculated in impairment percentages, with higher numbers indicating greater impaired quality of life.

CONTACTS AND LOCATIONS:
Locations (2):
- CLINUVEL Investigational site, Clinuvel Investigational Site, Belgium
- CLINUVEL Investigational site, Clinuvel Investigational Site, Spain